CLINICAL TRIAL: NCT02957591
Title: The Effect of Probiotic Supplementation on the Efficacy of Antidepressant Treatment in Depression
Brief Title: Probiotic Supplementation in Severe Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Principal Investigator, André Schmidt, Ph.D., Psychiatric Hospital of the University of Basel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-01608
Record Dates: First submitted 2016-11-01; First posted 2016-11-08 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Severe Depression
Keywords: Depression; probiotic supplementation; Adjuvant Therapy; Gut microbiome; Psychological functioning; Brain imaging; Brain-Gut interactions; Sleep
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Over a period of 4 weeks, depressive patients will ingest a probiotic food supplementation (Vivomixx®) 4 times a day. Primary and secondary endpoints will be assessed before and after the intervention.
  Interventions: Dietary Supplement: Vivomixx®
- Placebo Group (Placebo Comparator): Subjects in the placebo group will receive a placebo 4 times a day over 4 weeks. Primary and secondary endpoints will be assessed before and after the intervention.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx® — Streptococcus thermophilus Bifidobacterium breve Bifidobacterium longum Bifidobacterium infantis Lactobacillus acidophilus Lactobacillus plantarum Lactobacillus paracasei Lactobacillus delbrueckii subsp. bulgaricus
  Arms: Probiotic Group
Other: Placebo — Subjects in the placebo group will receive a placebo that contains starch but no bacteria. The appearance of the placebo will be indistinguishable in color, shape, size, packaging, smell, and taste from that of the probiotic supplement.
  Arms: Placebo Group

SUMMARY:
Recent research demonstrates that the composition of the gut microbiome is a master regulator of key neurophysiological processes that are affected in depression. Indeed, contemporary studies showed that faecal microbiota is altered in patients with major depressive disorder (MDD). Furthermore, it has also been shown that supplementation of probiotics ameliorated depressive symptoms in unmedicated patients with mild to moderate depression. However, no study has yet explored the efficacy of a probiotic-based therapy in patients with severe MDD in addition to a standard antidepressant treatment. As dietary and lifestyle interventions may be a desirable, effective, pragmatical and non-stigmatizing prevention and adjuvant therapy (in addition to antidepressant treatment) in depression, this project is aimed at investigating for the first time if probiotic supplementation compared to a placebo treatment improves the effect of standard antidepressant medication on depressive symptoms (i.e. better and faster remission) in patients with severe MDD. Furthermore, this study will further test if probiotic supplementation modulates immune signalling and inflammatory processes (macrophage migration inhibitory factor and interleukin 1 beta), hypothalamic-pituitaryadrenal (HPA) axis responses (saliva cortisol), neurogenesis (brain-derived neurotrophic factor (BDNF) expression), the release of appetite-regulating hormones (leptin and ghrelin), the composition of gut microbiota (in particular levels of Enterobacteriaceae, Alistipes and Faecalibacterium) and brain perfusion, structure and activation and if these changes are associated with the probiotic-induced effect on depressive symptoms.

DETAILED DESCRIPTION:
Major depression is a recurrent and debilitating mental disorder with a lifetime prevalence of up to 20% in the general population, among the highest for psychiatric disorders. Its diagnosis is based upon the presence of persisting affective, cognitive and behavioural symptoms, with a depressive episode requiring at least five of these symptoms during a period of at least two weeks. When considering the biological mechanisms that underpin depression, the most conclusive findings include deficits in the serotonergic (5-HT) neurotransmission, alterations in the expression of BDNF, deficient immune activation and neuroinflammation, and dysregulation of the hypothalamic-pituitary-adrenal (HPA) axis. Thus, understanding the pathophysiological mechanisms of MDD has widespread implications for the development of novel treatment and prevention strategies. However, despite advancements in the development of novel therapeutics, current treatment options have not reached optimal efficacy. Treatment resistant depression occurs in up to 40% of patients and standard antidepressant medication has a variety of undesirable side effects such as sedation, decrease of blood pressure, increase of weight, indigestion or sexual dysfunction. This often results in patients' poor compliance resulting in a break-up of medication with recurrence of depressive symptoms and increased suicidal risk. As there is an unmet need to develop safer and more effective treatments in depression, a major topic of future psychiatric care is to focus on different possible physiologically relevant mechanisms in order to establish alternative, causative and easy available treatment strategies.

In the past few years, it has become increasingly evident that resident gut bacteria are an important contributor to healthy metabolism and there is significant evidence linking altered composition of the gut microbiota and metabolic disorders such as obesity and depression. Preclinical work in animals have reported associations between alterations of the gut microbiome (the community of microorganism that live in the human gut) and anxiety-like behaviour, depressive-like symptoms and stress responsiveness. In line with these preclinical findings, a recent study found an altered composition of faecal microbiota in patients with MDD. Most notably, the MDD group had increased levels of Enterobacteriaceae and Alistipes but reduced levels of Faecalibacterium, which was negatively correlated with the severity of depressive symptoms.

Accumulating evidence suggest that there exits a bi-directional communication system between the gastrointestinal tract and the brain. Changes in gut microbiota can influence cognitive and emotional stress processes through interactions with the brain and altered emotional states and dysfunction of the gut microbiome-brain axis has been implicated in stress-related disorders such as depression. Brain-gut interactions could occur in various ways: 1) microbial compounds communicate via the vagus nerve, which connects the brain and the digestive tract, and 2) microbially derived metabolites interact with the immune system, which maintains its own communication with the brain. Although the pathways linking gut bacteria with the brain are incompletely understood, one of the principal mechanisms proposed to underlie stress-induced alterations is the "leaky gut" phenomenon. Specifically, increased translocation of bacterial products, due to a compromised gut barrier has been linked to activation of the immune system and HPA axis. In line with these findings, human studies have demonstrated a stress-induced increase in bacterial translocation in depression. The stress-induced interactions between the gut microbiome and the brain are further mediated via central processes such as neurotransmission and neurogenesis. For instance, there is substantial evidence to demonstrate a role for the gut commensals in the regulation and development of the 5-HT system and the expression of BDNF. Virtually all corticolimbic brain structures that are involved in mood regulation and stress response express 5-HT receptors. These include the prefrontal cortex, amygdala, hippocampus and nucleus accumbens. A recent meta-analyses of fMRI studies support hyperactivation of several of these regions in response to fearful faces in MDD, which extent correlated positively with the severity of depressive symptoms. Furthermore, during resting state fMRI, MDD patients showed lower connectivity between the amydgala, hippocampus, parahippocampus, and brainstem, while the connectivity strength was inversely correlated with general depression. The hippocampus, and its connection to other limbic, striatal and PFC regions, seems to play a key role in stress regulation, given that hippocampal neurogenesis mediates antidepressant effects via the ventral hippocampus' influence on the HPA axis, and mechanisms by which antidepressants may reverse chronic stress-induced 5-HT and neurogenic changes. Notably, BDNF may contribute to the modulation of neurogenesis in response to both stress and antidepressants, as hippocampal BDNF levels decrease in response to chronic stress and increase in response to antidepressant treatments.

Besides being a fundamental player in eating processes and in hypothalamic regulation of energy balance, the appetite-regulating hormones leptin and ghrelin had been implicated in the etiology of mood disorders. Importantly, particular species of bacteria in the gut are know to affect the levels of leptin and ghrelin. In humans, the onset of depression was associated with a combination of high leptin levels coupled with high visceral fat, and the link between leptin levels and severity of depressive symptoms was mediated by adiposity. It was suggested that leptin might influence depression by acting on leptin receptors present on 5-HT neurons within the raphe nuclei and dopamine neurons in the midbrain and, thus, might influence reward processes. Consistent with this supposition, when leptin receptors in the rat hippocampus were genetically deleted, a stressor-induced depressive profile was apparent, and deletion of leptin receptors on midbrain dopamine neurons in mice elicited elevated anxiety. Thus, identifying the key brain regions that mediate leptin's antidepressant activity and dissecting its intracellular signal transduction pathways may provide new insights into the pathogenesis of depression and facilitate the development of novel therapeutic strategies for the treatment of this illness.

The gut peptide ghrelin also plays a fundamental role in eating and energy regulation and there have been indications that ghrelin functioning might contribute to depressive illness. Like leptin, ghrelin receptors have been reported in the midbrain and the dorsal raphe nucleus and have been associated with reward processes, as well as stressor-induced depressive-like symptoms, such as anhedonia. In line with a role for ghrelin in stressor-elicited depression, negative events promote an increase of circulating ghrelin levels and in emotionally reactive individuals the normalization of ghrelin levels after stress may be attenuated. Moreover, ghrelin was elevated among depressed patients and declined following pharmacotherapy and among patients who did not respond to treatment, ghrelin levels were higher than among patients who responded positively.

Compelling preclinical data demonstrated the beneficial effect of probiotics in normalizing HPA axis functioning, BDNF levels and 5-HT neurotransmission. In particular, certain probiotics such as lactobacilli and bifidobacteria can reverse psychological stress-induced HPA axis activation and possess antidepressant or anxiolytic activity in rats. A seminal work in experimental animals showed that altered stress responsiveness has been partially reversed by colonization of the gut. Importantly, a recent and innovative study showed that short-term consumption of mostly animal or mostly plant diet rapidly and reproducibly altered the human gut microbiome, suggesting that the development of dietary interventions may provide a novel promising adjuvant therapy in addition to pharmacological antidepressant treatments in MDD. Indeed, recent reports of trials administrating a combination of probiotics to healthy subjects demonstrated improvements in depression or anxiety outcome measures. Moreover, urinary free cortisol levels were significantly reduced by the probiotics, providing a potential mechanism for the improvement in psychological symptoms observed. Consistent with this finding, other studies in healthy subjects found that the consumption of a probiotic-containing yogurt improved mood and that a multispecies probiotic (different strains of lactobacilli and bifidobacteria) reduced rumination and aggressive thoughts. Moreover, a pioneer study in healthy subjects revealed by using fMRI that consumption of probiotic bacteria (including strains of lactobacilli and bifidobacteria) in fermented milk for 4 weeks modulated brain activation in corticolimbic regions while viewing frightened and angry facial expressions. Most important, a very recent study demonstrated that administration of probiotics, a mixture of lactobacilli and bifidobacteria, ameliorated depressive symptoms in unmedicated patients with mild to moderate depression. These studies together suggest that restoring disturbed gut microbiome-brain interactions via probiotic bacteria might be a desirable treatment strategy for depression, especially as most of the clinically depressed patients additionally suffer from obesity, weight loss or gain, appetite disturbances and constipation.

This project is aimed at investigating for the first time if probiotic supplementation improves the effect of antidepressants on depressive symptoms (i.e. better and faster remission) in patients with severe MDD. Furthermore, this study will also test if probiotic supplementation modulates immune signalling and inflammatory processes, HPA axis responses, neurogenesis, the release of appetite-regulating hormones, the composition of gut microbiota and brain perfusion, structure and activation and if these changes are associated with the probiotic-induced effect on depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18.
* Mild depression (Hamilton Depression Rating Scale (HAM-D) > 7).
* Inpatient with antidepressant treatment at the UPK Basel.
* Treatment as usual for depression

Exclusion Criteria:

* Comorbid psychiatric disturbances such as substance abuse disorder, bipolar disorder, schizophrenia.
* Current medical conditions such as acute infectious disease, dietary restrictions.
* Immunosuppressed patients
* Pregnancy, breast-feeding.
* Inability to read and understand the participant's information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Score | Change from baseline at week four

SECONDARY OUTCOMES:
Brain perfusion | Change from baseline at week four
  measured with arterial spin labeling (ASL)
Brain structure | Change from baseline at week four
  measured with diffusion tensor Imaging (DTI)
Brain activation | Change from baseline at week four
  measured with functional magnetic resonance imaging (fMRI)
HPA axis function | Change from baseline at week four
  measured with salivary cortisol awakening responses
Neurogenesis | Change from baseline at week four
  measured with blood levels of BDNF
Appetite-regulating hormones | Change from baseline at week four
  measured with blood levels of ghrelin and leptin
Immunoregulation and inflammation | Change from baseline at week four
  measured with blood levels of macrophage migration inhibitory factor and interleukin 1 beta
Beck depression score | Change from baseline at week four
Psychopathology | Change from baseline at week four
  measured with the Brief Symptom Check List (BSCL)
Cognition | Change from baseline at week four
  measured with the Trail Making Test A and B
State and trait anxiety | Change from baseline at week four
  measured wit the State-Trait Anxiety Inventory (STAI)
Social interactions | Change from baseline at week four
  measured with the Reading the Mind in the Eyes task
Physical activity | Change from baseline at week four
  measured with the International physical activity questionnaire (IPAQ) and Fitbit-Flex®, a portable wristwatch
Sleep quality | Change from baseline at week four
  measured with 3-channel electroencephalography (EEG) and the Insomnia Severity Index
Gut microbiota composition | Change from baseline at week four
  via faecal sampling
Gastrointestinal side effects | Change from baseline at week four

CONTACTS AND LOCATIONS:
Overall Officials: André Schmidt, Ph.D., Principal Investigator — University Psychiatric Clinics (UPK); Laura Mählmann, M.Sc., Principal Investigator — University Psychiatric Clinics (UPK); Stefan Borgwardt, Professor, Principal Investigator — University Psychiatric Clinics (UPK)
Locations (1):
- University Psychiatric Clinics (UPK), Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sempach L, Doll JPK, Limbach V, Marzetta F, Schaub AC, Schneider E, Kettelhack C, Mahlmann L, Schweinfurth-Keck N, Ibberson M, Lang UE, Schmidt A. Examining immune-inflammatory mechanisms of probiotic supplementation in depression: secondary findings from a randomized clinical trial. Transl Psychiatry. 2024 Jul 24;14(1):305. doi: 10.1038/s41398-024-03030-7. PMID 39048549
- [Derived] Schneider E, Doll JPK, Schweinfurth N, Kettelhack C, Schaub AC, Yamanbaeva G, Varghese N, Mahlmann L, Brand S, Eckert A, Borgwardt S, Lang UE, Schmidt A. Effect of short-term, high-dose probiotic supplementation on cognition, related brain functions and BDNF in patients with depression: a secondary analysis of a randomized controlled trial. J Psychiatry Neurosci. 2023 Jan 18;48(1):E23-E33. doi: 10.1503/jpn.220117. Print 2023 Jan-Feb. PMID 36653035
- [Derived] Schaub AC, Schneider E, Vazquez-Castellanos JF, Schweinfurth N, Kettelhack C, Doll JPK, Yamanbaeva G, Mahlmann L, Brand S, Beglinger C, Borgwardt S, Raes J, Schmidt A, Lang UE. Clinical, gut microbial and neural effects of a probiotic add-on therapy in depressed patients: a randomized controlled trial. Transl Psychiatry. 2022 Jun 3;12(1):227. doi: 10.1038/s41398-022-01977-z. PMID 35654766